CLINICAL TRIAL: NCT03401619
Title: Beijing Osteoporosis With Neurological Disorders in Epigenetic Changes Study: an Ambispective, Multicentre, Open Cohort Study
Brief Title: Beijing Osteoporosis With Neurological Disorders in Epigenetic Changes Study
Acronym: BONE
Status: Active, not recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Ministry of Education, China (Other Government); Beijing Municipal Science & Technology Commission (Other); Ministry of Science and Technology of the People´s Republic of China (Other Government); Peking University Health Science Center (Other)
Responsible Party: Principal Investigator, Dongwei Fan, Orthopeadic doctor, Peking University Third Hospital
Other Study IDs: BONEM2017294
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Last update posted 2020-09-17 (Actual); Status verified 2020-09

CONDITIONS: Osteoporosis，Neurological Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Osteoporosis With Cognitive impairment
  Interventions: Combination Product: Exercise，Nutrition，Bisphosphonates，Statins，Calcitonin,Vitamin D，et al.
- Osteoporosis With Arterial stiffness
  Interventions: Combination Product: Exercise，Nutrition，Bisphosphonates，Statins，Calcitonin,Vitamin D，et al.
- Osteoporosis
  Interventions: Combination Product: Exercise，Nutrition，Bisphosphonates，Statins，Calcitonin,Vitamin D，et al.
- Normal
  Interventions: Combination Product: Exercise，Nutrition，Bisphosphonates，Statins，Calcitonin,Vitamin D，et al.

INTERVENTIONS:
Combination Product: Exercise，Nutrition，Bisphosphonates，Statins，Calcitonin,Vitamin D，et al. — The long-term effect of comprehensive treatment on health, especially for osteoporosis and neurodegenerative diseases, we hope to find association from epigenetics and provide clues for further exploration of its pathogenesis.

SUMMARY:
Epigenetic modification refers to the change of heritable gene expression occurring in the case of unchanged DNA sequence, including DNA methylation, epigenetic modification, RNAS, chromatin modification, etc. The study found that osteoporosis (OSTEOPOROSIS,OP) with neurological disorders is very common, the risk of fracture of patients increased. It is considered that epigenetic regulation plays an important role in the occurrence and development of OP with neurological disorders. In particular, the role and molecular mechanism of epigenetic modification in OP with neurological disorders are not clear, and the results of clinical studies with different sample sizes are not consistent. (1) Two-way continuous queues,an ambispective cohort study， namely: forward-looking queue method (2017-2027) and Retrospective queue method (2007-2017) were used to understand the effect of epigenetic modification on bone mineral density, bone metabolic Biochemical Index, imaging index and fracture incidence of patients with neurological diseases in outpatients and wards, and to provide basis for further study. To observe the effects of epigenetic modification on cognitive function in two groups of patients (memory scale, life activity Energy meter (ADL) and cognitive scale (MMSE) and clinical physical examination and neuropsychological test, etc., Bone correlation detection (Lumbar and hip bone mineral density T-score, imaging index, bone Metabolic Biochemical Index and fracture incidence index) Influence. Multivariate stepwise regression analysis was performed to eliminate confounding factors, such as age, body mass index (BMI), related risk factors, and internal diseases. The patient's previous information is also analyzed; (2) To find meaningful epigenetic modification from clinical data, the molecular mechanism was studied in depth, and the imaging indexes (X-ray, CT, MRI) and Bone marker Index (serum osteocalcin (OC), total I-type procollagen peptide (TP1NP) were found in the study. Type I collagen hydroxy-terminated peptide beta degradation product (Β-CTX)). The relationship between the reaction epigenetic modification and cognitive function index, image and bone markers and the mechanism model were further established.

ELIGIBILITY:
Inclusion Criteria:

* Normal hearing, vision, and pronunciation
* DEXA examination

Exclusion Criteria:

* Mental retardation
* Blindness, deafness, and dumb
* Severe schizophrenia

Ages: 55 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer, outpatient, inpatient
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-09-21 (Actual); Primary Completion 2026-09-22 (Estimated); Study Completion 2027-09-22 (Estimated)

PRIMARY OUTCOMES:
cognitive impairment improvement | year 1,2,3,4 and 5
  Change from baseline in Mild Cognitive Impairment assessment scale-cognitive subscale in year 1,2,3,4 and 5

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Dubois B, Feldman HH, Jacova C, Hampel H, Molinuevo JL, Blennow K, DeKosky ST, Gauthier S, Selkoe D, Bateman R, Cappa S, Crutch S, Engelborghs S, Frisoni GB, Fox NC, Galasko D, Habert MO, Jicha GA, Nordberg A, Pasquier F, Rabinovici G, Robert P, Rowe C, Salloway S, Sarazin M, Epelbaum S, de Souza LC, Vellas B, Visser PJ, Schneider L, Stern Y, Scheltens P, Cummings JL. Advancing research diagnostic criteria for Alzheimer's disease: the IWG-2 criteria. Lancet Neurol. 2014 Jun;13(6):614-29. doi: 10.1016/S1474-4422(14)70090-0. PMID 24849862
- [Background] Norton S, Matthews FE, Barnes DE, Yaffe K, Brayne C. Potential for primary prevention of Alzheimer's disease: an analysis of population-based data. Lancet Neurol. 2014 Aug;13(8):788-94. doi: 10.1016/S1474-4422(14)70136-X. PMID 25030513
- [Background] Vos SJ, Xiong C, Visser PJ, Jasielec MS, Hassenstab J, Grant EA, Cairns NJ, Morris JC, Holtzman DM, Fagan AM. Preclinical Alzheimer's disease and its outcome: a longitudinal cohort study. Lancet Neurol. 2013 Oct;12(10):957-65. doi: 10.1016/S1474-4422(13)70194-7. Epub 2013 Sep 4. PMID 24012374
- [Background] Barnes DE, Yaffe K. The projected effect of risk factor reduction on Alzheimer's disease prevalence. Lancet Neurol. 2011 Sep;10(9):819-28. doi: 10.1016/S1474-4422(11)70072-2. Epub 2011 Jul 19. PMID 21775213
- [Background] Villemagne VL, Burnham S, Bourgeat P, Brown B, Ellis KA, Salvado O, Szoeke C, Macaulay SL, Martins R, Maruff P, Ames D, Rowe CC, Masters CL; Australian Imaging Biomarkers and Lifestyle (AIBL) Research Group. Amyloid beta deposition, neurodegeneration, and cognitive decline in sporadic Alzheimer's disease: a prospective cohort study. Lancet Neurol. 2013 Apr;12(4):357-67. doi: 10.1016/S1474-4422(13)70044-9. Epub 2013 Mar 8. PMID 23477989
- [Background] Wilkinson D, Windfeld K, Colding-Jorgensen E. Safety and efficacy of idalopirdine, a 5-HT6 receptor antagonist, in patients with moderate Alzheimer's disease (LADDER): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2014 Nov;13(11):1092-1099. doi: 10.1016/S1474-4422(14)70198-X. Epub 2014 Oct 5. PMID 25297016
- [Background] Leder BZ, Tsai JN, Uihlein AV, Wallace PM, Lee H, Neer RM, Burnett-Bowie SA. Denosumab and teriparatide transitions in postmenopausal osteoporosis (the DATA-Switch study): extension of a randomised controlled trial. Lancet. 2015 Sep 19;386(9999):1147-55. doi: 10.1016/S0140-6736(15)61120-5. Epub 2015 Jul 2. PMID 26144908
- [Background] Sestak I, Singh S, Cuzick J, Blake GM, Patel R, Gossiel F, Coleman R, Dowsett M, Forbes JF, Howell A, Eastell R. Changes in bone mineral density at 3 years in postmenopausal women receiving anastrozole and risedronate in the IBIS-II bone substudy: an international, double-blind, randomised, placebo-controlled trial. Lancet Oncol. 2014 Dec;15(13):1460-1468. doi: 10.1016/S1470-2045(14)71035-6. Epub 2014 Nov 11. PMID 25456365

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-09-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03401619/SAP_000.pdf